CLINICAL TRIAL: NCT07335640
Title: Impact d'Une Fiche Explicative donnée Aux Parents après Une première Consultation Pour Crise fébrile Simple au Service d'Accueil Des Urgences pédiatriques du CHU de Strasbourg
Brief Title: Impact of an Information Sheet Given to Parents After an Initial Consultation for a Simple Febrile Seizure at Strasbourg University Hospital
Acronym: ConvulStop
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9695
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Febrile Crisis
Keywords: Febrile crisis; Simple febrile crisis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Simple febrile seizures (SFS) are a very common phenomenon (2-5% of children), mostly without serious consequences for the child or their development, but extremely anxiety-provoking for parents, who develop a "fear of fever" for fear of a recurrence, and request numerous additional tests, not justified according to current guidelines, after a first episode of SFS.

Educating parents about these fever-related crises and fever management, and standardizing the information provided through an explanatory sheet implemented at the SAUP in July 2023, would help reduce consultations for recurrent simple febrile crises, as well as early consultations for isolated fever (reflecting parental anxiety caused by these crises).

ELIGIBILITY:
Inclusion Criteria:

* Child aged between 9 months and 5 years at the time of consultation at the SAUP (emergency pediatric unit)
* First visit to the SAUP for a simple febrile seizure
* Meeting the clinical criteria for FCS:

  * Generalized seizure lasting less than 15 minutes
  * No post-critical deficit
  * No recurrence of seizures within 24 hours
  * No personal history of neurological disorders
* Occurrence between January 1, 2022, and May 1, 2025
* First or second episode of FSFS at the time of consultation
* Presence of one of the two parents during the consultation at the SAUP

Exclusion Criteria:

* Patient already seen at the SAUP for FCS
* Child who has already had more than two simple febrile seizures at the time of their visit to the emergency department.
* Child who does not meet the criteria for simple febrile seizures:
* aged less than 9 months or more than 5 years at the time of diagnosis.
* Non-febrile seizure
* Focal seizure
* Seizure duration >15 min
* Presence of post-critical deficit
* Multiple seizures within 24 hours
* Personal neurological history.
* Seizure occurring outside the period of interest (January 1, 2022 to May 1, 2025)
* Absence of parents during the SAUP consultation

Ages: 9 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: - Child aged between 9 months and 5 years at the time of consultation at the SAUP (emergency pediatric unit)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Number of consultations at the Pediatric Emergency Department for recurrent simple febrile crises. | Up to 4 years
  Number of consultations at the Pediatric Emergency Department (SAUP) for recurrent simple febrile crises.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France